CLINICAL TRIAL: NCT04005378
Title: Disengagement in CSC: Identifying Those at Risk and Addressing Their Needs
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-0307 -B
Record Dates: First submitted 2019-07-01; First posted 2019-07-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: First Episode Psychosis

STUDY DESIGN:
Intervention Model Description: Assigned to either treatment as usual or to the disengagement treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSC Step-down intervention (Other): Web-based telemedicine and a smartphone app, to decrease disengagement likelihood
  Interventions: Other: CSC Step-down intervention
- Usual Care (Other): Usual care provided by CSC center
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: CSC Step-down intervention — Web-based telemedicine and a smartphone app, to decrease disengagement likelihood
  Arms: CSC Step-down intervention
Other: Usual Care — Usual Care provided by CSC center
  Arms: Usual Care

SUMMARY:
Maintaining treatment engagement is critical for first episode psychosis patients to experience gains possible with coordinated specialty care (CSC). This study is designed to identify CSC participants still receiving care but at high risk for disengagement and to intervene to prevent/delay disengagement.

DETAILED DESCRIPTION:
In Phase 1 of the project, we will confirm a model predicting factors associated with later disengagement from CSC treatment. In Phase 2, we will compare disengagement among high-risk individuals with a CSC Step-down intervention to that with standard CSC care. The Step-down intervention will use web-based telemedicine and a smartphone app, to decrease disengagement likelihood. High-risk participants identified by predictors found in Phase 1 will be offered the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled into a CSC program

Exclusion Criteria:

* None

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Disengagement rate | Minimum of 6 months
  Rate of disengagement from CSC program

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Henderson Behavioral Health, Lauderdale Lakes, Florida
  - InterAct of Michigan, Grand Rapids, Michigan
  - InterAct of Michigan, Kalamazoo, Michigan

IPD SHARING:
Plan to Share IPD: No